CLINICAL TRIAL: NCT01555060
Title: Hemoglobin and Iron Recovery Study
Acronym: HEIRS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Institute for Transfusion Medicine (Unknown); Versiti Blood Health (Other); Blood Centers of the Pacific (Unknown); American National Red Cross (Other); University of California, San Francisco (Other); Vitalant Research Institute (Other); RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 714
Record Dates: First submitted 2012-03-09; First posted 2012-03-15 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Recovery of Hemoglobin and Iron Stores After Blood Donation
Keywords: hemoglobin recovery; iron recovery; iron supplements
MeSH Terms: interventions — ferrous gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iron supplements (Experimental): Subjects who are randomized to receive daily iron supplements after donating blood
  Interventions: Dietary Supplement: ferrous gluconate
- Control (No Intervention): Subjects who are randomized not to receive daily iron supplements after donating blood

INTERVENTIONS:
Dietary Supplement: ferrous gluconate — daily capsule of ferrous gluconate containing 38 mg of elemental iron
  Arms: Iron supplements

SUMMARY:
The purpose of this study is to investigate the effect of daily iron supplements after blood donation on time to recovery of hemoglobin and iron stores. The study will also determine whether the effect of iron supplements on time to recovery is different in men and women, in older vs. younger donors (<60 years old vs. at least 60 years old) and in donors with replete vs. diminished pre-donation iron stores.

DETAILED DESCRIPTION:
The effect of taking iron supplements after blood donation on time to recovery of hemoglobin has been documented but it is not clear whether the benefits of iron supplements vary with age, gender or iron stores. To study this issue, individuals who are eligible to donate blood, based on hemoglobin level, will be randomized to receive daily iron supplements or no supplements. Randomization will be stratified on gender (male or female), age (<60 years old vs. at least 60 years old) and iron status (serum ferritin >26 vs serum ferritin no greater than 26). Subjects will be followed for 24 weeks with periodic blood draws to determine time to recovery of hemoglobin and iron stores. A 7 ml (about 1.5 teaspoons) blood sample will be drawn at each of seven study visits over the 24 weeks to track recovery of hemoglobin and iron.

ELIGIBILITY:
Inclusion Criteria:

* potential blood donors with hemoglobin of at least 12.5 gm/dL
* no blood donation for at least 4 months
* successful donation of a unit of whole blood

Exclusion Criteria:

* individuals who are taking iron supplements including multivitamins containing iron and refuse to stop do so for the 24 weeks of the study.
* baseline ferritin >300 ug/L (to exclude individuals with hemochromatosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Time to recovery of hemoglobin after blood donation | Up to 24 weeks after blood donation
  Hemoglobin will be measured 3-7 days and 2, 4, 8, 12, 16 and 24 weeks after blood donation. A nonlinear regression of hemoglobin vs time since donation will be used to determine time to recovery of hemoglobin to 80% of the pre-donation level.

SECONDARY OUTCOMES:
Iron stores | Up to 24 weeks after blood donation
  Ferritin will be measured 3-7 days and 2, 4, 8, 12, 16 and 24 weeks after blood donation. A nonlinear regression of hemoglobin vs time since donation will be used to determine time to recovery of to pre-donation iron stores.
Total body iron | 24 weeks after blood donation
  Soluble transferrin receptor (sTfR) in blood will be measured 3-7 days and 24 weeks after blood donation. The ratio of sTfR to ferritin will provide a measure of total body iron at the two time points. Recovery of total body iron will be estimated from the difference between the ratios at the two time points.

CONTACTS AND LOCATIONS:
Overall Officials: Joe Kiss, MD, Principal Investigator — Institute for Transfusion Medicine
Locations (4):
- United States (4):
  - Blood Centers of the Pacific, San Francisco, California
  - American Red Cross, Connecticut Region, Farmington, Connecticut
  - Institute for Transfusion Medicine, Pittsburgh, Pennsylvania
  - Blood Center of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Mast AE, Szabo A, Stone M, Cable RG, Spencer BR, Kiss JE; NHLBI Recipient Epidemiology Donor Evaluation Study (REDS)-III. The benefits of iron supplementation following blood donation vary with baseline iron status. Am J Hematol. 2020 Jul;95(7):784-791. doi: 10.1002/ajh.25800. Epub 2020 Apr 15. PMID 32243609
- [Derived] Cable RG, Brambilla D, Glynn SA, Kleinman S, Mast AE, Spencer BR, Stone M, Kiss JE; National Heart, Lung, and Blood Institute Recipient Epidemiology and Donor Evaluation Study-III (REDS-III). Effect of iron supplementation on iron stores and total body iron after whole blood donation. Transfusion. 2016 Aug;56(8):2005-12. doi: 10.1111/trf.13659. Epub 2016 May 27. PMID 27232535
- [Derived] Kiss JE, Brambilla D, Glynn SA, Mast AE, Spencer BR, Stone M, Kleinman SH, Cable RG; National Heart, Lung, and Blood Institute (NHLBI) Recipient Epidemiology and Donor Evaluation Study-III (REDS-III). Oral iron supplementation after blood donation: a randomized clinical trial. JAMA. 2015 Feb 10;313(6):575-83. doi: 10.1001/jama.2015.119. PMID 25668261